CLINICAL TRIAL: NCT06906874
Title: Efficacy and Safety of Activated Charcoal on Mineral Bone Disorder in Chronic Kidney Disease Patients
Brief Title: Activated Charcoal Use in Chronic Kidney Disease Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha Mansour, Principal investigator-Associate Professor of Clinical Pharmacy-Clinical Pharmacy and Pharmacy Practice Department, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-117'2
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease (ESRD); CKD 5D, Hemodialysis; CKD-MBD - Chronic Kidney Disease Mineral and Bone Disorder
MeSH Terms: conditions — Kidney Failure, Chronic; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — Charcoal

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Other): patients receiving standard care therapy of calcium-based or non-calcium based (sevelamer) binders.
  Interventions: Drug: Phosphate Binders
- Intervention group (Experimental): patients receiving standard care therapy of calcium-based or non-calcium based (sevelamer) binders in addition to oral activated charcoal capsules with meals
  Interventions: Drug: Activated Charcoal; Drug: Phosphate Binders

INTERVENTIONS:
Drug: Activated Charcoal — oral activated charcoal capsules
  Arms: Intervention group
Drug: Phosphate Binders — calcium-based or non-calcium based (sevelamer) binders

SUMMARY:
Hyperphosphatemia management is initially based on restricting dietary phosphorus intake. Hyperphosphatemia is almost always seen in patients on dialysis and may contribute to progressive vascular calcification. Considering that activated charcoal is generally well-tolerated and may have a favorable side effect profile compared to conventional phosphate binders, it presents a promising alternative. Until now, no clinical trial has primarily investigated the effect of activated charcoal on hyperphosphatemia in dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged ≥18 years with ESRD.
2. Patients who had been on stable maintenance hemodialysis (3 times weekly) for at least 6 months.
3. Patients receiving phosphate binders according to standard protocols established by kidney disease: Improving Global Outcomes (KDIGO).

Exclusion Criteria:

1. Severely malnourished (as diagnosed by the department's dietitian).
2. Treated with overnight dialysis.
3. Primary hyperparathyroidism or persistent serum levels of intact parathyroid hormone greater than 800 pg/mL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Serum phosphorus levels | 8 weeks
  Difference between two groups of serum phosphorous level in mg/dL at the end of the study.

SECONDARY OUTCOMES:
The percentage of patients who achieved decreasing at least 3 points in The Worst Itching Intensity Numerical Rating Scale (WI NRS) | 8 weeks
  The (WI-NRS) is a validated 11-point scale, with scores ranging from 0 to 10 and with higher scores indicating greater itch intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Please Select, Egypt